CLINICAL TRIAL: NCT04776395
Title: Iberdomide in Intermediate- and High-Risk Smoldering Myeloma (SMM) Patients: A Phase 2 Study With a Safety Run-in
Brief Title: Iberdomide Alone or in Combination With Dexamethasone for the Treatment of Intermediate- or High-Risk Smoldering Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nisha Joseph, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001731; NCI-2020-08351 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP5157-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-03-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (iberdomide hydrochloride, dexamethasone) (Experimental): Patients receive iberdomide hydrochloride PO QD on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive iberdomide hydrochloride PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Iberdomide Hydrochloride; Other: Quality-of-Life Assessment
- Arm B (iberdomide hydrochloride) (Active Comparator): Patients receive iberdomide hydrochloride PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Iberdomide Hydrochloride; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Iberdomide Hydrochloride — Given PO
  Other Names: CC-220 Hydrochloride
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the effects of iberdomide when given alone or in combination with dexamethasone in treating intermediate or high-risk smoldering multiple myeloma patients. Immunotherapy with iberdomide may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread. Dexamethasone is a synthetic steroid (similar to steroid hormones produced naturally in the adrenal gland), and is used with other drugs in the treatment of some types of cancer. Giving iberdomide with dexamethasone my improve time to progression to symptomatic myeloma with improved tolerability.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) of iberdomide hydrochloride (iberdomide) and iberdomide with dexamethasone in intermediate- and high-risk smoldering multiple myeloma (SMM).

SECONDARY OBJECTIVES:

I. To determine the 1- and 2- year progression free survival rates of patients receiving iberdomide with and without dexamethasone in intermediate-risk and high-risk smoldering myeloma.

II. To determine the time to progression, and overall survival of patients with intermediate- and high-risk smoldering myeloma receiving iberdomide with and without dexamethasone.

III. To study the risk of adverse hematologic and non-hematologic events observed in patients receiving iberdomide with and without dexamethasone for treatment of intermediate- and high-risk smoldering myeloma.

IV. To evaluate stem cell mobilization failure and early stem cell mobilization feasibility.

TERTIARY/EXPLORATORY OBJECTIVES:

I. To assess the effects of iberdomide on cereblon targets Aiolos and Ikaros in natural killer (NK)- and T- cells.

II. To measure the effect of iberdomide with and without dexamethasone on T-cell and NK-cell counts and activation.

III. To determine the prognostic impact of high-risk cytogenetic abnormalities on clinical outcomes.

IV. To assess minimal residual disease (MRD) on bone marrow samples in subjects who achieved a complete response (CR) or better and evaluate the correlation between MRD status and clinical outcome measures.

V. To assess the association between anti-tumor activity and immune cells in tumor and blood.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive iberdomide hydrochloride orally (PO) once daily (QD) on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive iberdomide hydrochloride PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive iberdomide hydrochloride PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have intermediate- or high risk smoldering multiple myeloma (SMM) as confirmed by at least one of the following factors either at screening or within 28 days of screening:

  * Bone marrow clonal plasma cells >= 20% confirmed on either screening bone marrow biopsy or by outside pathology ≤5 years from initiation of study drug.
  * Abnormal serum free light chain ratio > 20 by serum free light chain (FLC) assay
  * Serum monoclonal protein >= 2 g/dL
* Subject must have been diagnosed with SMM =< 5 years from initiation of study drug
* Both men and women of all races and ethnic groups are eligible for this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky >= 60%) is required for eligibility
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin (Hgb) > 11 g/dL
* Platelet count >= 100,000 cells/mm^3 and must be platelet and packed red blood cells (PRBC) transfusion independent with no granulocyte colony-stimulating factor (G-CSF) to ensure eligibility within 8 weeks of screening
* Estimated creatinine clearance >= 30 mL/min as defined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) or Cockcroft-Gault
* Total bilirubin < 2 mg/dL except in subjects with congenital bilirubinemia such as Gilbert syndrome, in which case direct bilirubin =< 2 times the institutional upper limit of normal is required
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times the institutional upper limit of normal
* Left ventricular ejection fraction >= 40%
* Females of childbearing potential (FCBP) must have two negative pregnancy tests as verified by the investigator prior to starting study treatment. The effects of Iberdomide on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact. A FCBP must either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of iberdomide. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Female of childbearing potential (FCBP) is a sexually mature woman who:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* The subject must be willing to comply with fertility requirements as below:

  * Male subjects must agree to use an adequate method of contraception for the duration of the study and for 3 months afterwards
  * Female subjects must be either postmenopausal, free from menses >= 2 years (yrs), surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from heterosexual activity starting with screening and for 3 months after last treatment in all patients
  * Patients must agree not to donate blood, sperm/ova while taking protocol therapy and for at least 4 weeks after stopping treatment
* Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* Multiple myeloma requiring treatment as defined by SLiM-CRAB criteria
* Monoclonal gammopathy of undetermined significance (MGUS), polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS syndrome), plasma cell leukemia, primary systemic light chain (AL) amyloidosis, or Waldenstroms macroglobulinemia
* Concurrent intravenous bisphosphonate use more often than once a year
* Prior or ongoing treatment for plasma cell disorder
* Active hepatitis B or C due to risk of infection made worse by study drug
* If subject has human immunodeficiency virus (HIV), they must have a CD4 count >= 350, no history of acquired immune deficiency syndrome-related illness, and not currently prescribed zidovudine or stavudine
* Subjects may be receiving concomitant low dose corticosteroids (e.g., prednisone up to but no more than 10 mg by mouth daily or its equivalent) for symptom management and comorbid conditions
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the preceding 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects with gastrointestinal disease that may significantly alter the absorption of iberdomide
* Pregnant women are excluded from this study because protocol therapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to protocol treatment of the mother, breastfeeding should be discontinued
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of iberdomide. The following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection); systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisone or equivalent steroids as premedication for hypersensitivity reactions (e.g, computed tomography [CT] scan pre-medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 3 years
  Assessed per International Myeloma Working Group response criteria (to be done with serum and urine immunologic studies monthly; bone marrow biopsy and repeat imaging at either complete response or progressive disease).

SECONDARY OUTCOMES:
Progression-free survival | From start of protocol therapy to disease progression or death from any cause, whichever comes first, assessed at 1 and 2 years
  Will be estimated with the Kaplan-Meier method with 95% confidence interval (CI) for the two randomized arms separately and combined. Cox proportional hazards models will be further used to compare the two randomized arm with hazard ratio and its 95% CI reported.
Time to progression | From start of protocol therapy to disease progression, assessed at 1 and 2 years
  Will be estimated with the Kaplan-Meier method with 95% CI for the two randomized arms separately and combined. Cox proportional hazards models will be further used to compare the two randomized arm with hazard ratio and its 95% CI reported.
Overall survival | From start of protocol therapy to death, censoring patients who are alive at last follow-up, assessed at 1 and 2 years
  Will be estimated with the Kaplan-Meier method with 95% CI for the two randomized arms separately and combined. Cox proportional hazards models will be further used to compare the two randomized arm with hazard ratio and its 95% CI reported.
Rate of grade 3-4 adverse events | Up to 30 days after the last day of study participation
  Adverse event data will be described and graded per the National Cancer Institute Common Terminology Criteria for Adverse Events guidelines. Grade 3-4 adverse events will be estimated as frequency and percentage, and then compared between the two patient groups using Chi-Square test.
Successful stem cell mobilization | Up to 3 years
  Defined as collection of 3.5 x 10^6 CD34 cells per kilogram weight.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha S Joseph, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States